CLINICAL TRIAL: NCT04746118
Title: Effectiveness of Nutritional Intervention Alone or Associated With Other Non-pharmacological Interventions in Controlling Hypertension and Reducing Cardiovascular Risk - Randomized Clinical Trial
Brief Title: Diet and Other Non Pharmacological Interventions to Reduce Cardiovascular Risk in Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitário Clementino Fraga Filho (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, ELIZABETH SILAID MUXFELDT, Medical Doctor, Hospital Universitário Clementino Fraga Filho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41740720.7.1001.5257
Record Dates: First submitted 2021-01-26; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: Resistant hypertension; Diet changes; Regular physical activity; Integrative practices; Pre-hypertension
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — Exercise; Auriculotherapy

STUDY DESIGN:
Intervention Model Description: Besides the control group (n=60), three other groups with different severity of hypertension will be included in the study. To evaluate strategies adopted as primary prevention 60 pre-hypertensive patients will be recruited. To evaluate blood pressure control and cardiovascular risk reduction, other 60 hypertensives will be also invited to the study. Finally, 60 individuals with resistant hypertension will be recruited to access secondary and tertiary prevention with possible blood pressure control, reduction in the number of drugs in use and subclinical lesions regression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CONTROL (No Intervention): During routine clinical visits the patients will receive a written standard general guidelines for diet and physical activity.
- DIET CHANGE (Experimental): In scheduled nutritional care the patients will receive an individual program with social media supervision. Those patients will also receive a written general guidelines for exercising without supervision.
  Interventions: Behavioral: DIET CHANGE
- DIET CHANGE + PHYSICAL ACTIVITY (Experimental): In scheduled nutritional care the patients will receive an individual program with social media supervision. Those patients will also receive an exercise physical program prescription with fitness evaluation and close supervision.
  Interventions: Behavioral: DIET CHANGE; Behavioral: PHYSICAL ACTIVITY
- DIET CHANGE + PHYSICAL ACTIVITY + INTEGRATIVE PRACTICES (Experimental): In scheduled nutritional care the patients will receive an individual program with social media supervision. Those patients will also receive an exercise physical program prescription with fitness evaluation and close supervision and submitted to orientated mind-fullness, auriculotherapy and "laying on of hands" approaches that belong to health integrative practices.
  Interventions: Behavioral: DIET CHANGE; Behavioral: PHYSICAL ACTIVITY; Other: INTEGRATIVE PRACTICES

INTERVENTIONS:
Behavioral: DIET CHANGE — Nutritional supervision will be carried out individually based on the Food Guide for the Brazilian Population, ensuring an accessible, hygienic and contextualized diet according to the subject's culture and physiology. The protocol includes an initial assessment to define the meal plan and individual reassessments every four weeks. In the first evaluation participants will receive an eating plan with a 20% reduction in the total calories consumed or even the equivalent of their daily energy needs with a distribution of macronutrients comprised of 65% carbohydrate, 15% protein and 20% fat. The intention is to promote a reduction in weekly consumption by about 2000 kilocalories (Kcal). The prescription and diet control plan will include and be conducted by a team coordinated by a clinical nutritionist.
  Other Names: Nutritional intervention
  Arms: DIET CHANGE; DIET CHANGE + PHYSICAL ACTIVITY; DIET CHANGE + PHYSICAL ACTIVITY + INTEGRATIVE PRACTICES
Behavioral: PHYSICAL ACTIVITY — The physical activity program will consist of daily walking sessions performed outdoors and on a flat surface suitable for hiking. Each session will last 70 minutes and will be performed between 55% -60% of the maximum oxygen consumption (VO2), six times a week, for 24 weeks, with alternate on-site supervision on odd days and remote monitoring on even days. On-site supervision will be carried out by a team coordinated by a Physical Education teacher and implemented at two times in the morning and another two in the afternoon with meeting points previously defined. At the end of each supervised walking session, 20 minutes of exercise will be performed using the equipment available at the Senior Citizens Academy set up in public squares in the region so that the total expenditure of calories spent weekly with physical activities reach about 2000 kilocalories.
  Other Names: Aerobic training and mobility exercises
  Arms: DIET CHANGE + PHYSICAL ACTIVITY; DIET CHANGE + PHYSICAL ACTIVITY + INTEGRATIVE PRACTICES
Other: INTEGRATIVE PRACTICES — The health integrative practices will includes Mind-Fullness, auriculotherapy and laying on of hands. A suitably qualified professional, using it use a practical manual so that the practice became uniform among the subjects, will apply the practice of Mind-Fullness in weekly 1-hour sessions to individuals. The practice of auriculotherapy will be applied to individuals by a professional qualified to perform the technique, which consists in the selection of auricular points according to the health problems presented and the therapeutic objectives that are to be achieved, followed by the insertion of the mustard seed at specific points in the ear over a six-month period. The laying on of hands will be carried out by properly trained individuals.
  Other Names: Holistic Health Integrative practices: mind-fullness meditation and auriculotherapy
  Arms: DIET CHANGE + PHYSICAL ACTIVITY + INTEGRATIVE PRACTICES

SUMMARY:
The purpose of this study is to evaluate the effectiveness of diet change and other non-pharmacological treatments which includes physical activity and integrative therapies oriented to reduce the blood pressure in hypertensive patients.

DETAILED DESCRIPTION:
Despite advances in the pharmaceutical industry, blood pressure control remains the biggest challenge in the treatment of hypertension in Brazil and worldwide. In this context, besides the availability and use of antihypertensive drugs, the best therapeutic approach should start with the stratification of cardiovascular risk, and contextualized modification of life habits. In this view, the present study aims to evaluate the effectiveness of diet change and other non-pharmacological treatments oriented to reduce the blood pressure in adults diagnosed with prehypertension, hypertension, and resistant hypertension. Therefore, it includes the analysis of these 3 groups: i. pre-hypertension (to evaluate strategies adopted as primary prevention); ii. hypertension in general (to assess blood pressure control and reduce cardiovascular risk reduction), and iii. resistant hypertension (individuals using 3 or more drugs without blood pressure control who have more endothelial dysfunction and target organ damage to assess secondary and tertiary prevention with possible blood pressure control, reduction in the number of drugs in use and subclinical lesions regression). Non-pharmacological approach includes adoption of healthy lifestyles, weight loss, reduced sodium intake, regular physical activity, and integrative practices capable of maintaining biopsychosocial balance. Since those interventions seems to be the best way to reach blood pressure control, we intend to use individual interventions and group actions to increase the population's adherence contributing effectively to public policies within primary care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes aged between 20 and 65 years old;
* Resistant hypertensive individuals: hypertensive individuals using 3 antihypertensive drugs or more without control of office blood pressure (BP ≥ 140 x 90 mmHg) or using 4 drugs with pressure control in follow-up at Hypertension Program (ProHArt) - University Hospital (HUCFF) - Federal University of Rio de Janeiro (UFRJ).
* Pre-hypertensive individuals: individuals with systolic blood pressure (SBP) between 121-139 mmHg and / or diastolic blood pressure (DBP) between 81-89 mmHg without the use of antihypertensive drugs registered at Family Health Strategy unit.
* Hypertensive: individuals with SBP ≥ 140 mmHg and / or DBP ≥ 90 mmHg or using antihypertensive drugs registered at Family Health Strategy unit.
* Individuals who accept to participate in the research after signing the Free and Informed Consent Form

Exclusion Criteria:

* Pregnant;
* Major cardiovascular events (acute myocardial infarction, unstable angina, stroke) in the last 6 months;
* Individuals with psychiatric illnesses or significant cognitive impairment;
* Individuals with clinical conditions that preclude physical activity such as severe peripheral arterial disease, advanced osteoarticular disease, neurological degenerative disease, severe muscle disease;
* Individuals who have undergone weight loss procedures (diet or medication) in the last 6 months;
* Individuals who have undergone surgical procedures for weight loss;
* Individuals who are participating in any other intervention study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 21 months
  Indicators: Office blood pressure and Home Blood Pressure Monitoring (HBPM) after 6 months of non-pharmacological intervention Goals: Nutritional strategy: reduction of 1 mmHg by reducing each kg of body weight and reducing salt intake reaching <1.5 g / day with a reduction of 2 to 3 mmHg.
  Physical activity: reduction of 6 to 8 mmHg in office systolic blood pressure and 4 to 6 mmHg in HBPM with good adherence to moderate aerobic exercise Integrative practices: 4 mmHg reduction in systolic blood pressure

SECONDARY OUTCOMES:
Body weight | 21 months
  Indicators: Body weight reduction after 6 months of non-pharmacological intervention Goals: reduction of body weight by 0.9 kg to 1.1 kg each month It is believed that the nutritional intervention and physical activity group has a higher monthly weight loss, reaching up to 2 kg / month.
Body composition | 21 months
  Indicators: the reduction in fat mass is expected in all intervention groups with an increase in lean muscle mass, especially in groups 2 and 3, which include physical activity. The goal is to achieve a lean mass of over 30% in women and 33% in men.

OTHER OUTCOMES:
Glycidic profile | 21 months
  Indicators: laboratory tests - glycated hemoglobin after 6 months of non-pharmacological intervention Goals: Glycated hemoglobin reduction <6,0%
Lipidic profile | 21 months
  Indicators: laboratory tests - lipogram after 6 months of non-pharmacological intervention Goals: Total cholesterol < 200 mg/d
Triglycerides | 21 months
  Indicators: laboratory tests - serum triglycerides after 6 months of non-pharmacological intervention Goals: triglycerides < 150 mg/dL
Left ventricular hypertrophy | 21 months
  Indicators: ECG voltage indices (left ventricular hypertrophy) reduction after 6 months of non-pharmacological intervention.
  Goals: Reduction of Sokolow-Lyon index (SV1 + RV5)
Renal function | 21 months
  Indicators: glomerular filtration rate (GFR) after 6 months of non-pharmacological intervention Goals: Increase GFR > 60 ml/min/m2 body surface area (BSA)
Albuminuria | 21 months
  Indicators: albuminuria in urinary spot Goals: Reduction of Albuminuria < 30mg/g creatinine
Aortic stiffness | 21 months
  Indicators: pulse wave velocity (PWV) measurement (aortic stiffness) Goals: reduction of aortic stiffness measured by PWV < 10 m/s
Endothelial dysfunction | 21 months
  Indicators: Laser Doppler flowmetry (microvascular reactivity reflects endothelial dysfunction) Goals: increase microvascular reactivity with a percentage > 10%
Improved quality of life | 21 months
  Indicators: scores obtained in the World Health Organization Quality of Life questionnaire (WHOQOL-Bref) Goals: Improvement of the 4 domains investigated in the WHOQOL-Bref: physical health, psychological, social relationships and environment.
  Results in % varies from 0 to 100. The higher the percentage (closer to 100%) the better the quality of life.
Obstructive Sleep Apnea (OSA) risk | 21 months
  Indicators: scores obtained in the Stop-Bang (Snoring, Tiredness, Observed apnea, high blood Pressure, Body mass index, Age, Neck circumference, and Gender) questionnaires indicate high risk for OSA:- STOP-BANG score > 3 Goals: Reduce the STOP-BANG score to <3
Excessive daytime sleepiness | 21 months
  Indicators: scores obtained in the Epworth Sleepiness Scale (ESS) indicate excessive sleepiness and possible high risk for OSA: (ESS > 10.) Goals: Reduce the ESS score to <10.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth S. Muxfeldt, PhD Dr., Principal Investigator — Hospital Universitário Clementino Fraga Filho
Locations (1):
- Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Schwingshackl L, Chaimani A, Hoffmann G, Schwedhelm C, Boeing H. Impact of different dietary approaches on blood pressure in hypertensive and prehypertensive patients: protocol for a systematic review and network meta-analysis. BMJ Open. 2017 Apr 26;7(4):e014736. doi: 10.1136/bmjopen-2016-014736. PMID 28446526
- [Background] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Background] Lopes S, Mesquita-Bastos J, Alves AJ, Ribeiro F. Exercise as a tool for hypertension and resistant hypertension management: current insights. Integr Blood Press Control. 2018 Sep 20;11:65-71. doi: 10.2147/IBPC.S136028. eCollection 2018. PMID 30288097